CLINICAL TRIAL: NCT05861583
Title: Evaluation of Lipoedema Tissue Transcriptome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Schleswig-Holstein (Other)
Collaborators: Hanse-Klinik, Fachklinik für Liposuktion, Lübeck (Unknown); Praxisklinik Kronshagen, Kiel-Kronshagen (Unknown)
Responsible Party: Principal Investigator, Tobias Kisch, Principal Investigator, University Hospital Schleswig-Holstein
Other Study IDs: Lipo2023
Record Dates: First submitted 2023-05-06; First posted 2023-05-17 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Lipedema
Keywords: lipoedema; transcriptomics; fat tissue
MeSH Terms: conditions — Lipedema

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Lipohypertrophy: Active Comparator Tissue from healthy patients with lipohypertrophy,
  Interventions: Other: fat tissue
- Lipoedema mild stage: Experimental Tissue from lipoedema patients with mild stage (stage 1)
  Interventions: Other: lipoedema tissue (stage 1)
- Lipoedema moderate stage: Experimental Tissue from lipoedema patients with moderate stage (stage 2)
  Interventions: Other: lipoedema tissue (stage 2)
- Lipoedema severe stage: Experimental Tissue from lipoedema patients with severe stage (stage 3)
  Interventions: Other: lipoedema tissue (stage 3)

INTERVENTIONS:
Other: fat tissue — fat tissue sample collected while cosmetical liposuction
  Groups: Lipohypertrophy
Other: lipoedema tissue (stage 1) — lipoedema tissue sample (stage 1) collected while medical liposuction
  Groups: Lipoedema mild stage
Other: lipoedema tissue (stage 2) — lipoedema tissue sample (stage 2) collected while medical liposuction
  Groups: Lipoedema moderate stage
Other: lipoedema tissue (stage 3) — lipoedema tissue sample (stage 3) collected while medical liposuction
  Groups: Lipoedema severe stage

SUMMARY:
Lipoedema is a chronic painful disease with a fat distribution disorder affecting women. It is probably aggravated by hormonal changes. It is also discussed that a genetical predisposition might be a risk factor for developing lipoedema. The mechanisms leading to lipoedema are mostly unknown. The aim of this study is to identify molecular mechanisms and changes of the RNA-Expression pattern causing lipoedema by comparing the transcriptome of subcutaneous tissue of lipoedema patients vs. healthy subcutaneous tissue.

DETAILED DESCRIPTION:
Lipoedema is a fat distribution disorder affecting mostly women. This chronic disease is characterized by painful fatty tissue accumulating especially at the limbs. The aetiopathogenesis of this disease is unsure. It is observed that a familial predisposition might increase the risk of developing lipoedema. Hormonal variations during puberty, pregnancy or climacteric period are also discussed as main factor for lipoedema. Molecular and genetical changes are rarely identified. The aim of this study is to identify changes in the expression pattern of fat cells causing lipoedema. One possibility to medicate this disease is to reduce the subcutaneous fatty tissue by liposuction. While this surgical procedure, a tumescent solution for reducing bleeding and pain is used. This study is also trying to identify the effect of tumescent solution to fatty tissue.

This trial is an explorative study using excised tissue by surgery to compare the gene expression pattern of subcutaneous tissue of lipoedema patients to healthy subcutaneous tissue. Therefore, lipoedema patients of mild stage, moderate stage and severe stage as well as healthy patients with lipohypertrophy as control group are included to the study. The participation was on a voluntary basis. Only patients who reached the age of majority and who are able to consent were included.

The study group patients are characterized by the typical, symmetrical and painful fat distribution especially at the limbs. The aim of the surgical treatment via liposuction of lipoedema patients is to reduce the fatty tissue, which is causing the development of oedema, the persistent pain and the formation of haematoma. The control group patients are determined by having a healthy subcutaneous fatty tissue, which was surgical reduced caused by cosmetical effects. The subcutaneous tissue therefore was reduced via liposuction following the standardised operation procedures. Starting the procedure, a small native tissue sample is collected without any additional invasive procedure. After installing a tumescent anaesthetic solution containing epinephrine and local anaesthetics subcutaneous the liposuction will be performed. The liposuction is done in power assisted liposuction technique. An additional sample of liposuctioned fat tissue treated with tumescent solution will be collected. The RNA-Expression pattern of the fatty tissue will be analysed by performing a NGS-Analysis. Changes of the RNA-Expression of lipoedema of different stages compared to normal fatty tissue will be detected. Further the effect of the intra-surgical used tumescent solution on fat cells can be detected by comparing native and treated tissue samples.

Another aim of the study is to collect data concerning anamnestic aspects, symptoms and factors possibly leading to the development and progress of the disease. These data will be analysed to identify risk factors for lipoedema.

ELIGIBILITY:
Inclusion Criteria:

1. Lipohypertrophy: tissue from healthy patients (n=20): Consent-capable female patients ≥18 years of age with lipohypertrophy
2. Lipoedema milde stage: tissue from Lipoedema patients with mild stage 1 (n=20): Consent-capable female patients ≥18 years of age with Lipoedema (Stage 1)
3. Lipoedema moderate stage: tissue from Lipoedema patients with moderate stage 2 (n=20): Consent-capable female patients ≥18 years of age with Lipoedema (Stage 2)
4. Lipoedema severe stage: tissue from Lipoedema patients with severe stage 3 (n=20): Consent-capable female patients ≥18 years of age with Lipoedema (Stage 3)

Exclusion Criteria:

* Inflammation in region of interest, HIV, Hepatitis

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Consent-capable female patients ≥18 years of age with either lipohypertrophy or lipoedema
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Differences in RNA-Expression pattern | 1 day
  Differences in RNA-Expression pattern between lipoedema tissue and lipohypertrophy tissue

CONTACTS AND LOCATIONS:
Locations (1):
- University of Schleswig-Holstein, Lübeck, Schleswig-Holstein, Germany

REFERENCES:
- [Derived] Streubel MK, Baumgartner A, Meier-Vollrath I, Frambach Y, Brandenburger M, Kisch T. Transcriptomics of Subcutaneous Tissue of Lipedema Identified Differentially Expressed Genes Involved in Adipogenesis, Inflammation, and Pain. Plast Reconstr Surg Glob Open. 2024 Nov 8;12(11):e6288. doi: 10.1097/GOX.0000000000006288. eCollection 2024 Nov. PMID 39525887